CLINICAL TRIAL: NCT05937659
Title: Incorporating Biometric Data Evaluation for Patients Receiving Concurrent Chemotherapy and Radiation Therapy
Brief Title: Incorporating Biometric Data for Patients Receiving Concurrent Chemotherapy & RT
Status: Not yet recruiting | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: LCCC2237
Record Dates: First submitted 2023-06-30; First posted 2023-07-10 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Cancer
Keywords: radiation therapy; chemotherapy; biometric data; wearable health technology
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Biometric Data Collection: Adult subjects with cancer and prescribed concurrent systemic therapy and radiation therapy and enrolled in the study.

SUMMARY:
This study will assess the feasibility of incorporating biometric data via wearable health technology (WHT) into the radiation oncology (RO) clinic workflow for patients receiving concurrent radiation therapy and systemic therapy (CRT) for cancer. The investigators hypothesize that a practical workflow could be created within a busy community RO practice that will allow providers and patients to readily appreciate physiologic declines during concurrent CRT.

Subjects will be asked to wear a device as part of this study that will collect their biometric data (heart rate, number of steps taken per day, etc) called a WHT device throughout their treatment and for 4 weeks afterward. Subjects will be asked to upload the data from their devices onto the computers in the clinic for the assessment.

ELIGIBILITY:
Inclusion Criteria In order to participate in this study a subject must meet all of the eligibility criteria outlined below.

Subjects

1. All genders aged ≥ 18 years of age.
2. English-speakers
3. Able to understand and cooperate with study procedures.
4. Signed and dated informed consent.
5. Subjects being seen at Novant-New Hanover Regional Medical Center for diagnosis and management of cancer.
6. Subjects prescribed to receive concurrent radiation therapy and systemic therapy either definitively or postoperatively.
7. Signed and dated HIPAA authorization for the release of personal health information.

Providers

1. All genders aged ≥ 18 years of age.
2. English speakers.
3. Able to understand and cooperate with study procedures.
4. Signed and dated informed consent.

Exclusion Criteria Both Subjects and care providers

1. Has dementia, altered mental status, or any psychiatric or co-morbid condition prohibiting the understanding or rending of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult subjects were diagnosed with cancer and prescribed concurrent systemic therapy and radiation therapy and their providers.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-03-15 (Estimated); Primary Completion 2027-03-15 (Estimated); Study Completion 2027-03-15 (Estimated)

PRIMARY OUTCOMES:
The rate of technology adoption | Up to 12 weeks
  The rate of technology adoption will be quantified as the fraction of subjects who successfully download their WHT data into the research databases in the radiation oncology clinic. Success, on a subject-specific basis, will be defined as their reporting any of their WHT biometric data on >40% of eligible days.

SECONDARY OUTCOMES:
Provider perception of the utility | Up to 12 weeks
  The physician's and nurse's subjective assessment of the utility of having the subject's wearable health technology data such as enhanced dietary or hydration counseling, supportive medication alteration, and/or intravenous fluid hydration will be quantified, using a survey.
Subject perception of the utility | Up to 12 weeks
  The subjects' responses to the utility of wearable health technology data will be quantified using surveys.

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Mazur, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- Novant Health Cancer Institute Radiation Oncology, Wilmington, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No